CLINICAL TRIAL: NCT00923728
Title: A Phase 1 Trial of AVN944, an IMPDH Inhibitor, in Adults With Advanced Stage Solid Tumors
Brief Title: A Phase I Trial of AVN944, an IMPDH Inhibitor, in Adults With Advanced Stage Solid Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090119; 09-C-0119; NCT00890773 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2011-08

CONDITIONS: Refractory Solid Tumors
Keywords: AVN - 944; Phase I; Adult Solid Tumors; Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — AVN 944

INTERVENTIONS:
Drug: AVN944

SUMMARY:
Background:

* AVN944 is an experimental cancer treatment drug, not yet approved by the U.S. Food and Drug Administration. To date, AVN944 as a single drug has been tested in several studies involving humans, including healthy volunteers, patients with leukemia, and patients with advanced pancreatic cancer.
* More research is needed to determine the safety and effectiveness of AVN944.

Objectives:

* To determine the safety of AVN944.
* To determine the maximum tolerated dose (the highest dose that does not cause unacceptable side effects) of AVN944.
* To see if AVN944 has any effect on patients' tumors.
* To learn how the body breaks down AVN944.

Eligibility:

* Patients 18 years of age and older who have advanced stage solid tumors for which standard therapies do not exist or are no longer effective.

Design:

* Participants will have a screening visit and five clinic visits during the first treatment cycle. Additional treatment cycles will involve two clinic visits during each 28-day cycle. After participation in the study ends, patients will be asked to return within 28 days after the last dose of study drug for final study procedures.
* Evaluations before the treatment period:
* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Questions about medications and side effects.
* Blood and urine tests.
* Disease evaluation with CT, chest x-ray, and additional laboratory tests depending on the type of cancer.
* All patients will have blood samples taken at each visit.
* Patients will take specific doses of AVN994 as directed by researchers, and will be asked to keep a diary to record their doses and any side effects. They will be monitored with frequent blood draws at each study visit to provide information on the safety and effectiveness of the drug.
* During different cycles, patients will have their disease evaluated by researchers and will be asked if they wish to continue taking AVN994 as part of the study.

DETAILED DESCRIPTION:
Background:

* The rate limiting step in the synthesis of guanine nucleotides is catalyzed by the enzyme inosine monophosphate dehydrogenase (IMPDH) and so inhibition of this enzyme will result in depletion of guanine nucleotide pools, cessation of DNA synthesis, cell cycle block at the Gr(1)/S interface and interference with cell division.
* The reduction in guanine nucleotide pools interferes with the ability of G-coupled proteins to act as intracellular signal transducers. IMPDH inhibition.
* AVN944 is a small-molecule, uncompetitive inhibitor of cell proliferation.
* A Phase I study in patients with hematologic malignancies is active and accruing subjects. The maximum-tolerated dose (MTD) has not been reached and no pattern of organ-specific or dose-progressive toxicity has been observed.

Objectives:

Primary

* The dose limiting toxicities with AVN944 in patients with advanced stage solid tumors.
* The MTD with AVN944 in patients with advanced stage solid tumors.

Secondary:

* Pharmacokinetics and the pharmacodynamics of AVN944 by study cohort.
* The extent of IMPDH inhibition on tumor tissue and peripheral blood mononuclear cells (PBMC).
* The effect of AVN944 on tumors by measuring guanine nucleotide pools levels using PBMC's.
* The effect of AVN944 on tumors by analyzing expression of genes related to IMPDH.

Eligibility:

* Inclusion:

  * Patients must have histologically confirmed malignancy.
  * Patients must be at least 4 weeks since prior chemotherapy or radiation therapy and 2 weeks since prior hormonal therapy.
  * ECOG performance status less than or equal to 2.
  * Life expectancy of greater than 3 months.
  * Age greater than or equal to 18.
* Exclusion:

  * Patients with known active brain metastases or other CNS involvement.
  * History of allergic reactions attributed to compounds of similar chemical or biologic.
  * Prior treatment with an IMPDH-inhibitor.
  * History of solid organ transplant and are on IMPDFI inhibitors therapy.

Design:

* Phase I Trial using 3+3 trail design using starting cohort of 150 mg twice per day escalating to 750 mg twice per day.
* 60 patients to be enrolled over 30-36 months.
* AVN944 will be administered in 28 day treatment cycles.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histologically confirmed malignancy (histopathological documentation of cancer confirmed in the NCI Laboratory of Pathology at the National Institutes of Health, the Pathology Department at Walter Reed Medical Center, or the Pathology Department at National Naval Medical Center, prior to starting this study) that is metastatic or unresectable and for which standard therapies do not exist or are no longer effective.
2. Patients must be at least 4 weeks since prior chemotherapy or radiation therapy and 2 weeks since prior hormonal therapy except for gonadotropin releasing hormone (GnRH) analogues and any acute or serious side effects of those therapies should be Grade less than 1 or returned to baseline
3. Patients must be able and willing to take oral capsules.
4. ECOG performance status less than or equal to 2
5. Life expectancy of greater than 3 months
6. Patients must have acceptable organ and marrow function as defined below:

   * Leukocytes greater than or equal to 3,000/mcL
   * Absolute Neutrophil Count greater than or equal to 1,500/mcL
   * Platelets greater than or equal to 100,000/mcL
   * Total Bilirubin less than or equal to 1.5 times institutional ULN (patients with known Gilberts syndrome may have values as high as less than or equal to 3.0 X ULN)
   * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
   * Creatinine less than or equal to 1.5 times institutional upper limit of normal
7. The effects of AVN944 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Age greater than or equal to 18 Years. Because no dosing or adverse event data are currently available on the use of AVN944 in patients less than 18 years of age, children are excluded from this study.

EXCLUSION CRITERIA:

1. Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 14 days of the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication). Clinically significant toxicities from this therapy must have resolved to less than Grade 2.
2. Patients with known active brain metastases or other CNS involvement with less than 6 months since curative-intent treatment
3. Patients receiving growth factors
4. Prior treatment with an IMPDH-inhibitor e.g. Mycophenolate Mofetil, & Tiazofurin
5. Uncontrolled current illness requiring hospitalization or intravenous antibiotics within the past 7 days
6. Pregnant women are excluded from this study because AVN944 agent has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AVN944, breastfeeding should be discontinued if the mother is treated with AVN944.
7. History of solid organ transplant and are on IMPDH inhibitors (mycophenolate mofetil) therapy
8. HIV-positive patients
9. The following medications and/or treatments are not permitted during the trial (i.e., through completion of the post treatment follow-up) and would constitute exclusion from the protocol:

   * Any other investigational treatment
   * Any cytotoxic chemotherapy
   * Any other systemic anti-neoplastic therapy including, but not limited to, immunotherapy or monoclonal antibody therapy.
   * Any radiotherapy, including systemically administered radioisotopes.
   * Systemic corticosteroids.
   * Any hormonal therapy except GnRH agonists / antagonists for patients with prostate cancer or medroxyprogesterone
   * Growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
1. The dose limiting toxicities with AVN944 in patients with advanced stage solid tumors; 2. Maximum tolerated dose with AVN944 in patients with advanced stage solid tumors

SECONDARY OUTCOMES:
1. Single, repeat dose pharmacokinetics; 2. Inosine monophosphate dehydrogenase inhibition; 3. Anti-neoplastic responses

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sintchak MD, Fleming MA, Futer O, Raybuck SA, Chambers SP, Caron PR, Murcko MA, Wilson KP. Structure and mechanism of inosine monophosphate dehydrogenase in complex with the immunosuppressant mycophenolic acid. Cell. 1996 Jun 14;85(6):921-30. doi: 10.1016/s0092-8674(00)81275-1. PMID 8681386
- [Background] Allison AC, Hovi T, Watts RW, Webster AD. The role of de novo purine synthesis in lymphocyte transformation. Ciba Found Symp. 1977;(48):207-24. doi: 10.1002/9780470720301.ch13. PMID 415850
- [Background] Jackson RC, Weber G, Morris HP. IMP dehydrogenase, an enzyme linked with proliferation and malignancy. Nature. 1975 Jul 24;256(5515):331-3. doi: 10.1038/256331a0. No abstract available. PMID 167289